CLINICAL TRIAL: NCT02962193
Title: Evaluation of Functional and Social Changes After Bariatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Farraj Moaad, Dr, Western Galilee Hospital-Nahariya
Other Study IDs: 0043-16-NHR
Record Dates: First submitted 2016-11-06; First posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Functional and Social Performance
Keywords: ADL; Bariatric surgery; Daily participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
After bariatric surgery there are big changes in the daily functions, activities and social participation of the patients.

This is a prospective study that examine daily performance and daily participation by questionnaires, before and after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Overweight patients who are fit for surgery .

Exclusion Criteria:

* Children, Neurological patients, amputations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Overweight patients who are fit for surgery .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The change of participation before and after surgery | the patient will answer the questionnaire before and after (3 months, 6 months) surgery.

SECONDARY OUTCOMES:
sexuality questionnaire | the patient will answer the questionnaire before and after (3 months, 6 months) surgery.
activity daily questionnaire | the patient will answer the questionnaire before and after (3 months, 6 months) surgery.
range of motion (flexion of knee and thigh in degrees) | measure will be taken before and after (3 months, 6 months) surgery.
circumferences mesurement (knee, thigh and waist) in centimeters | measure will be taken before and after (3 months, 6 months) surgery.